CLINICAL TRIAL: NCT06555952
Title: MegaNatural BP® GSE on Blood Pressure and Cardiometabolic Risk Factors
Acronym: GSEBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024_081
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Pre Diabetes
MeSH Terms: conditions — Hypertension; Glucose Intolerance | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, 2-arm parallel, 6-week study
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GSE Capsule (Experimental): 150mg Grapeseed Extract MegaNatural BP
  Interventions: Dietary Supplement: MegaNatural-BP SR 150Mg Tablet
- Placebo Capsule (Placebo Comparator): Placebo supplement in place of GSE capsule
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: MegaNatural-BP SR 150Mg Tablet — GSE MegaNatural BP
  Arms: GSE Capsule
Other: Placebo Capsule — given in place of GSE MegaNatural BP
  Arms: Placebo Capsule

SUMMARY:
Inflammation and stressors can interfere with the function of the lining of blood vessels and insulin activity, therefore, investigators are aiming to see how the Grape seed Extract (GSE) called MegaNatural BP can help with limiting the effects of these factors. This research will study the effects of taking 150mg of MegaNatural BP GSE per day on blood pressure levels along with influences on heart health through assessing the function of the blood vessel lining and levels of inflammation.

DETAILED DESCRIPTION:
This is a research study to determine if an extract made from grape seeds might help control blood pressure. Previous research studies have found that taking this extract as a daily supplement at 300 mg per day in a capsule or a beverage may lower blood pressure in individuals with elevated blood pressure levels. The commercial name of this supplement is called MegaNatural BP®. The principal investigators of this study were part of the original research studies on GSE (both MegaNatural BP GSE and MegaNatural Gold GSE). They are now interested to determine if a lower amount of the grape seed extract might be effective in lowering people's blood pressure when its elevated. There is also some earlier information suggesting the GSE may influence how well insulin works in people's body. This may be helpful for individuals with metabolic conditions like the early stages of pre-diabetes.

The study will last for six weeks. All participants will visit the Clinical Nutrition Research Center (CNRC) seven times over the course of the study. These visits include a screening visit, two ambulatory blood pressure device fitting visits, and four study day visits throughout the six weeks. Blood will be collected to assess insulin activity measures during subject visits to the CNRC. The flexibility of subject's blood vessels will be measured using an ultrasound technique. Flexibility of vessels is important for blood pressure regulation and GSE has been known to help them become more flexible.

SCREENING VISIT

A subject's eligibility for the study is based on the list (inclusion and exclusion criteria). Clinical Research Coordinators will determine if the subject qualifies for the study at the Screening Visit by the following measurements:

* General measurements: height, weight, body composition and body temperature
* Fasting blood glucose from a finger prick
* Blood pressure
* Pregnancy test, for women under the age of 60 During the visit, the subject will be asked to complete a questionnaire or answer questions related to their health, dietary habits, and physical activity history. Based on the results of the blood sugar, questionnaires, measurements and evaluation of their health, the subject may meet the criteria and be invited to participate in the study.

PRE-STUDY / PRE-INTERVENTION VISIT (which may be performed at the same or different day as screening visit) The Pre-Study visit lasts ~30-45 minutes and the subject will meet with one of the investigators who will provide detailed instructions on procedures of the study (Blood pressure devices) and "how to prepare for each of the study days." The subject will be trained on all study procedures including, but not limited to foods to avoid during the study, medications/supplements to avoid, food diary recording, and GI-tract diary recording, fasting overnight. The participants study dates will be scheduled, and they will be provided a study booklet, including the study calendar and all instructions covered at the Pre-Study Visit.

Medications/Supplements: If the subject is taking any medications or supplements that do not interfere with the study or have been OK'd by study staff, they will take those as instructed by their doctor and will record in the diary. Clinical Research Coordinators will train the subject on what foods or supplements are OK and NOT OK during the study at the Pre-Study Visit.

Self-Characteristics and Dietary Surveys: During this visit, participants will be asked to complete online surveys that cover usual gastrointestinal (GI) symptoms and a 24-hour food recall.

Ambulatory Blood Pressure Device Fitting and Baseline BP measurement (Day 0) At the pre-study visit or another scheduled day at the participants convenience, the subject will be fitted with an ambulatory blood pressure device (ABPD) for collection of blood pressure for 24 h during their wake and sleep time. This is the most accurate assessment of their true blood pressure. They will begin wearing the device once fitted until returning the next day, which they will need to return to the clinic. As part of the 24 h device wearing, investigators will ask that the subject keeps a sleep, wake, exercise, eating diary. This helps the clinic understand the subject's data and when the blood pressure increases and decreases.

The subject will be given a frozen dinner to consume before they start fasting. This meal will be the same meal that is consumed before Visit 5.

STUDY DAY VISITS

Study Visit 1 / Day 1 Procedures

1. Staff collects study materials from participant

   1. Blood pressure monitor. Confirm data
   2. Diary and provide 24 h recall ASA24h
2. Confirmation the subject is ready to go for their study day by interview/discussion with study staff

   1. Fasted overnight for 10-12 hours
   2. Had a usual night of sleep
   3. Avoided alcohol and vigorous physical activity 24 hours before study day After confirming the subject is ready for their study day, staff will proceed to measure their weight, check their vital signs (blood pressure, heart rate and temperature) as well as measure their fasting blood glucose from a finger prick, ultrasound for FMD, body composition and collect a blood sample.

Ultrasound for Flow mediated dilation (FMD): FMD is a procedure to test the flexibility of brachial vessels. The researcher will use an ultrasound machine to visualize the artery in the subject's arm. The sonographer, who will visual the arm artery and conduct the procedure, will add sensors to the subject's body to track their heart rate and inflate a blood pressure cuff for 5 minutes on their arm before releasing to see and measure by ultrasound how flexible the arteries are. This will take about 30 minutes. The procedure will take place again 120 min after breakfast.

Blood collection: The subject will see the Licensed Health Care Provider (LHCP) for blood sample collection. The subject has the choice of an intravenous catheter or multiple butterfly sticks. There will be eight blood draws total. Once the fasting blood draw is collected, investigators will provide the subject with a capsule and then 5 min later a breakfast in the form of a nutritionally complete liquid drink (Ensure). Blood samples will be collected over the next 3 hours via a multi-sampling protocol. The subject will then be provided capsules for daily intake over two weeks until the next visit.

Other procedures. Every effort will be made to ensure the subjects safety while participating in this study.

Anthropometrics: Researchers will measure the subject's height as well as weight and body composition. Researchers will repeat the weight measurements as shown in the table. The subject will be asked to wear light comfortable clothing when coming to the screening and study related visits.

Vital signs: Researchers will check the subjects blood pressure, heart rate and body temperature using standard clinic devices.

Demographic questionnaire, health and medication questionnaire: Subjects will be asked to provide personal information, such as name, date of birth, race, etc. They will also be asked to answer questions about demographics, health, medical history, and the medications they take.

Study Visits 2 and 3 Procedures- Pick Up Visit Visit 2 (two weeks after Visit 1) and Visit 3 (two weeks after Visit 2) will involve a weight check, blood draw for compliance and supplement refill and reconciliation.

Study Visit 4- ABPD Fitting Procedure One day before Visit 5, the subject will be expected to come into the CNRC to be fitted with an ABPD. The subject will wear the ABPD day and night and fill out the 24 hour log until returning to the clinic for the final visit 5 the next day.

The subject will be given a frozen dinner to consume before they start fasting. This meal is the same as PreStudy or before Visit 1.

Study Visit 5 Procedures Visit 5 (two weeks after Visit 3) is the final study day visit. This visit will take place the day after Visit 4. This visit will be exactly the same as Visit 1, except the LMTT will include a capsule of the dietary regimens (placebo or MN-BP) that are randomly assigned to participants. After all study procedures are completed, the participant will be given a take-home snack and compensation will be issued.

ELIGIBILITY:
Inclusion Criteria:

* 40-60 years of age
* BMI < 30kg/m2
* elevated blood pressure 120-140 mmHg (systolic) / <90 mmHg (diastolic) at screening visit
* Has fasting blood glucose concentration between 100-125 mg/dL or HbA1c 5.7-6.4%.
* Not taking any medications that would interfere with outcomes of the study, i.e. blood pressure lowering medications or anti-diabetes medications.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study foods, records of food diary and GI tolerance questionnaire, sample collection procedures and study visit schedule)
* Able to maintain usual physical activity pattern
* Able to avoid / abstain from alcohol and vigorous physical activity for 24 hours prior to and during study visit

Exclusion Criteria:

* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or interventions
* Men and women with diabetes or have documented liver, kidney, cardiac, gastrointestinal, metabolic or respiratory diseases.
* Men and women with documented physical or mental disease/condition or major surgery as revealed by history or physical examination, which might limit participation in or completion of the study or, that, in the opinion of the investigator, could interfere with the interpretation of the study results.
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Taking medication or dietary supplements that may interfere with the outcomes of the study; This may include anti-inflammatory medication (ibuprofen, Aleve/naproxen, aspirin, etc.)
* Major trauma or a surgical event within 2 months (or longer depending on trauma or event) and after consultation with PI.
* Has used antibiotics within the previous 2 months
* Had colonoscopy within 3 months
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d)
* Donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours i.e., working overnight (e.g. 3rd shift)
* Follows a vegan diet or any extreme dietary patterns

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change of systolic blood pressure | 6 weeks
  After 6 weeks of 150mg GSE MegaNatural BP per day the base level blood pressure should change
Difference in change of diastolic blood pressure | 6 weeks
  After 6 weeks of 150mg GSE MegaNatural BP per day the base level blood pressure should change

SECONDARY OUTCOMES:
Change in vessel flexibility | 6 weeks
  Change in vessel flexibility as measured by flow mediated vasodilation acutely and chronically after GSE MegaNatural BP
Change in fasting and postprandial glucose | 6 weeks
  Change in fasting and postprandial glucose as measured by absolute values and calculated insulin sensitivity using homeostasis model assessment of fasting insulin senisitivity (HOMA-%S) and B-cell function (HOMA-%) and assessment of peripheral insulin sensitivity using Matsuda index.
Change in fasting and postprandial insulin | 6 weeks
  Change in fasting and postprandial insulin as measured by absolute values and calculated insulin sensitivity using homeostasis model assessment of fasting insulin senisitivity (HOMA-%S) and B-cell function (HOMA-%) and assessment of peripheral insulin sensitivity using Matsuda index.
Change in inflammatory marker C-reactive protein | 6 weeks
  additional plasma collected and saved for future analysis as study results warrant
Change in the ratio of arginine:ADMA | 6 weeks
  will be analyzed using High Performance Liquid Chromatography with mass analysis capabilities of mass spectrometry (MS)
Change in GSE metabolites profiles | 6 weeks
  will be analyzed using High Performance Liquid Chromatography with mass analysis capabilities of mass spectrometry (MS)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Principal Investigator — 708-563-8276
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No